CLINICAL TRIAL: NCT01031368
Title: Clofarabine in Combination With Cytarabine (Ara-C) and G-CSF Priming Followed by Infusion of Ex Vivo Expanded Cord Blood Progenitors for Patients With AML
Brief Title: Clofarabine, Cytarabine, and Filgrastim Followed by Infusion of Non-HLA Matched Ex Vivo Expanded Cord Blood Progenitors in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nohla Therapeutics, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2335.00; NCI-2009-01333 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Clofarabine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, G-CSF, cord blood infusion) (Experimental): INDUCTION THERAPY: Patients receive clofarabine IV over 1 hour and cytarabine hydrochloride IV over 2 hours on days 1-5. Patients receive an infusion of non-HLA matched ex vivo expanded cord blood progenitors on day 6. G-CSF is administered SC on days 0-5 and from day 7 until blood counts recover. Treatment modifications may apply according to response.
  CONSOLIDATION THERAPY: Patients receive clofarabine IV over 1 hour and cytarabine hydrochloride IV over 2 hours on days 1-5. Patients also receive G-CSF SC beginning on day 0 and continuing until blood counts recover.
  Interventions: Drug: cytarabine; Drug: clofarabine; Drug: filgrastim; Biological: Ex-vivo expanded cord blood progenitor cell infusion; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Drug: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: Ex-vivo expanded cord blood progenitor cell infusion — Undergo ex vivo-expanded cord blood progenitor cell infusion
  Other Names: Dilanubicel; NLA101
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the safety and potential efficacy of infusing non-human leukocyte antigen (HLA) matched ex vivo expanded cord blood progenitors following treatment with clofarabine and cytarabine for patients with acute myeloid leukemia (AML). The combination of clofarabine, cytarabine (Ara-C) and granulocyte colony-stimulating factor (G-CSF) has been tested in earlier studies for the treatment of acute myeloid leukemia. In these previous clinical trials, this combination of drugs has been shown to have an anti-leukemia effect. However, the combination of clofarabine and Ara-C is profoundly myelosuppressive and immunosuppressive causing periods of neutropenia potentially lasting more than three weeks. During this period, patients are at increased risk of infections that can result in an increased risk of death. G-CSF is a growth factor that is used to help the white blood cells recover more quickly, but even with G-CSF, the use of clofarabine and Ara-C is often limited by the need to take long breaks between treatments to allow blood counts to recover. In our lab we have developed a method of growing or "expanding" blood stem cells (cells that give rise to the blood system) from umbilical cord blood. We are doing this study to find out if giving these expanded cells after chemotherapy is safe, helps the blood system recover more quickly from chemotherapy to allow shorter breaks between treatments, and decreases the risk of infection

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of infusing off-the-shelf non-HLA matched expanded cord blood cells following administration of cytarabine hydrochloride (GCLAC) for patients with AML.

SECONDARY OBJECTIVES:

I. Assess the ability of the product to provide temporary myeloid engraftment.

II. Assess the kinetics/persistence of potential engraftment.

III. Assess the kinetics of autologous recovery when compared to historical cohorts.

IV. Assess the development of alloimmunization.

OUTLINE:

INDUCTION THERAPY: Patients receive clofarabine intravenously (IV) over 1 hour and cytarabine hydrochloride IV over 2 hours on days 1-5. Patients receive an infusion of non-HLA matched ex vivo expanded cord blood progenitors on day 6. Filgrastim (G-CSF) is administered subcutaneously (SC) on days 0-5 and from day 7 until blood counts recover. Treatment modifications may apply according to response.

CONSOLIDATION THERAPY: Patients receive clofarabine IV over 1 hour and cytarabine hydrochloride IV over 2 hours on days 1-5. Patients also receive G-CSF SC beginning on day 0 and continuing until blood counts recover.

Patients may receive treatment for 1-4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Diagnosis of AML by World Health Organization (WHO) criteria, either relapsed or refractory; acute promyelocytic leukemia [Acute promyelocytic leukemia with t(15;17)(q22;q12) and variants] will be eligible only after failure of a regimen containing arsenic trioxide; patients in this cohort must have had an initial remission duration of < 1 year and cannot have received any prior salvage chemotherapy
* Cohort B: Untreated AML patients, excluding those with favorable cytogenetic or molecular abnormalities per the European LeukemiaNet recommendations
* Cohort C: Untreated AML patients, including those with favorable cytogenetic or molecular abnormalities per the European LeukemiaNet recommendations
* The first three patients enrolled in cohorts A and B must be less than 60 years old; thereafter, patients aged >= 18 and =< 70 are eligible
* The first three patients enrolled in cohorts A and B must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 -1; thereafter, ECOG performance status of 0-2 is required
* Serum creatinine =< 1.0 mg/dL; if serum creatinine > 1.0 mg/dl, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation where predicted GFR (ml/min/1.73 m^2) = 186 X (Serum Creatinine)^-1.154 X (age in years)^-0.203 X (0.742 if patient is female) X (1.212 if patient is black)
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation is thought to be due to Gilbert's syndrome, hemolysis, or hepatic infiltration by the hematologic malignancy
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 X ULN, unless elevation is thought to be due to hepatic infiltration by the hematologic malignancy
* Alkaline phosphatase =< 2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must be willing to use an effective contraceptive method during the study and for a minimum of 90 days after study treatment

Exclusion Criteria:

* Allogeneic transplant recipients
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol with the exception of intrathecal chemotherapy administered on days that are not concurrent with clofarabine and cytarabine
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver (including symptomatic hepatitis, veno-occlusive disease), or other organ system dysfunction
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-10-24 (Actual)

PRIMARY OUTCOMES:
Grade 3 or greater infusion toxicity, as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 24 hours after expanded progenitor cell infusion
Treatment-related mortality | Up to 5 years
Platelet refractoriness in the presence of alloimmunization | Up to 6 months post-treatment
Exacerbation of chemotherapy-related toxicity, as defined by NCI CTCAE version 3.0 | Up to 21 days after initiation of clofarabine/cytarabine administration
Delayed marrow recovery (in the absence of relapse) when expanded cord blood progenitors are infused, defined as failure to achieve neutrophil recovery (ANC less than 500) post treatment with marrow cellularity and marrow blast count less than 5% | Up to day 35

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Delaney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Delaney C, Milano F, Cicconi L, Othus M, Becker PS, Sandhu V, Nicoud I, Dahlberg A, Bernstein ID, Appelbaum FR, Estey EH. Infusion of a non-HLA-matched ex-vivo expanded cord blood progenitor cell product after intensive acute myeloid leukaemia chemotherapy: a phase 1 trial. Lancet Haematol. 2016 Jul;3(7):e330-9. doi: 10.1016/S2352-3026(16)30023-0. Epub 2016 Jun 7. PMID 27374466